CLINICAL TRIAL: NCT06388993
Title: Comparison of the Constituents of Bone Marrow Aspirate and Autologous Protein Solution Collected With a Traditional and a Novel System
Brief Title: Marrow Cellution™ vs. Traditional BMA Harvest Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, William Vasileff, Associate Professor of Clinical Orthopedics, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023H0351
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hip Arthropathy; Avascular Necrosis of Bone; Subchondral Cysts
MeSH Terms: conditions — Osteonecrosis; Bone Cysts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Bilateral Hip Bone Marrow Collection (Experimental): Collection of bone marrow aspirate from both hips. One collected using the Zimmer Biomet Biocue system and the other using the Marrow Cellution system.
  Interventions: Device: Bone Marrow Collection

INTERVENTIONS:
Device: Bone Marrow Collection — Comparing the two collection systems for bone marrow aspirate

SUMMARY:
Six patients with diagnosed bone loss of the hip who have consented to minimally invasive repair will be approached to participate in the study. Participants will have the liquid portion of bone marrow collected using the Zimmer Biomet Biocue system, which is the standard system used by physicians at The Ohio State University, and the novel Marrow Cellutions system™. Bone marrow liquid will be collected from the surgical hip using the Zimmer Biomet Biocue system, and the Marrow Cellutions system™ will be used to collect bone marrow liquid from the non-surgical hip. Following collection, the bone marrow liquid will be processed using the respective systems to concentrate the cells and molecules found in the bone marrow liquid. As part of the standard of care for this arthroscopic procedure, concentrated bone marrow liquid processed using the Zimmer Biomet Biocue system will be delivered to the surgical site as an adjunct to promote healing. Concentrated bone marrow liquid prepared with the Zimmer Biomet Biocue system is given as part of the standard of care for patients undergoing minimally invasive treatment for bone loss of the hip; therefore, the target population for this study are individuals between the ages of 18-50 years with confirmed bone loss of the hip who have consented to minimally invasive repair. In addition to the concentrated bone marrow liquid prepared using the Zimmer Biomet Biocue system, patients will also have bone marrow liquid collected from the non-surgical hip using the Marrow Cellutions™ system. Only concentrated bone marrow liquid produced with the Zimmer Biomet Biocue system will be given to the patient. All concentrated bone marrow liquid produced with the Marrow Cellutions™ system will be sent to the laboratory for analysis. Additionally, white blood cells will be concentrated into an autologous protein solution (APS) using the Zimmer Biomet Plasmax system from blood collected using a routine blood draw. All protein solution produced will be sent to the laboratory for analysis. No protein solution will be given to the patient. As the bone marrow liquid collection using the Marrow Cellutions™ system and the blood draw to produce protein solution using the Zimmer Biomet Plasmax system are being performed for research,

DETAILED DESCRIPTION:
l

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 - 50
* patients undergoing hip arthroscopy for subchondral bone cysts and/or avascular necrosis

Exclusion Criteria:

* patients with a history of hematologic issues including anemia and sickle cell anemia
* patients with a history of leukemia, lymphoma, or other bone marrow related diseases
* patients with diabetes
* patients with a history of bone marrow aspirate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Assess overall number of stem cells collected from each aspiration method | 6 Months
  Compare total amount of stem cells collected from each sample

SECONDARY OUTCOMES:
Assess overall number of cytokines collected from each aspiration method | 6 Months
  Compare total amount of cytokines collected from each samples
Assess overall number of growth factors collected from each aspiration method | 6 Months
  Compare total amount of growth factors collected from each samples

CONTACTS AND LOCATIONS:
Overall Officials: William K Vasileff, MD, Principal Investigator — Ohio State University
Locations (1):
- Jameson Crane Sports Medicine Institute, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.